CLINICAL TRIAL: NCT04720742
Title: Immune Therapy and Analytical Treatment Interruption in HIV+ Participants Who Received an Allogeneic Stem Cell Transplantation (ITATI)
Brief Title: Immune Therapy and Analytical Treatment Interruption in HIV+ Participants Who Received an Allogeneic Stem Cell Transplantation
Acronym: ITATI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic the financial sponsor of the trial suspended the study funding due to funding limitations and based on various considerations, including the uncertainties of conducting the study in the volatile scenario of this pandemic.
Sponsor: IrsiCaixa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ITATI
Record Dates: First submitted 2019-12-12; First posted 2021-01-22 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: HIV Infection
Keywords: analytical treatment interruption; broadly neutralizing antibodies; immune therapy; allogeneic stem cell transplantation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: - Experimental group: the intervention will consist of an Analytical Treatment Interruption (ATI) of up to 18 months of duration, and during the first 8 months, a temporary immune intervention including the combination of the broadly neutralizing antibodies (bNAbs) 3BNC117 and 10-1074, which will be infused once per month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The participant will perform an Analytical Treatment Interruption (ATI) of up to 18 months of duration, and during the first 8 months, a temporary immune intervention including the combination of the broadly neutralizing antibodies (bNAbs) 3BNC117 and 10-1074, which will be infused once per month.
  Interventions: Drug: Analytical Treatment Interruption + bNAbs infusion

INTERVENTIONS:
Drug: Analytical Treatment Interruption + bNAbs infusion — The participant will perform an Analytical Treatment Interruption (ATI) of up to 18 months of duration. During the first 8 months, the participants will be infused once per month with a combination of the broadly neutralizing antibodies (bNAbs) 3BNC117 and 10-1074

SUMMARY:
The availability of antiretroviral therapy (cART) for HIV-1 infection has led to a reduction in morbidity in patients with chronic HIV infection. However, cART does not eliminate HIV-1 that persists as a latent infection in cellular reservoirs. Usually, HIV viremia rapidly rebounds if antiretroviral therapy is interrupted. Consequently, HIV infected individuals must commit to expensive, life-long therapies and must tackle problems associated with chronic infection and uninterrupted cART, including continuous clinical and laboratory monitoring, drug toxicities, and chronic immune activation/inflammation.

Currently, there is an emerging interest in developing safe and affordable curative strategies that would eliminate the need for lifelong therapy. However, to date only allogeneic hematopoietic stem cell transplantation (allo-HSCT) has shown results in decreasing the HIV-1 reservoirs.

The IciStem Consortium (www.icistem.org) has assembled the largest and most exhaustive observational cohort for the study of HIV reservoir dynamics in allo-HSCT HIV+ individuals with severe hematological malignancies worldwide. Within the cohort, only individuals transplanted with a donor with thw CCR5A32 mutation have shown signs of HIV remission. On the other side broadly neutralizing antibodies (bNAbs) have shown the potential to control HIV infection. This study intends to evaluate if the allo-HSCT combined with the additional application of bNAbs is effective to control HIV replication.

DETAILED DESCRIPTION:
The availability of antiretroviral therapy (cART) for HIV-1 infection has led to a reduction in morbidity in patients with chronic HIV infection. However, cART does not eliminate HIV-1 that persists as a latent infection in cellular reservoirs. Usually, HIV viremia rapidly rebounds if antiretroviral therapy is interrupted. Consequently, HIV infected individuals must commit to expensive, life-long therapies and must tackle problems associated with chronic infection and uninterrupted cART, including continuous clinical and laboratory monitoring, drug toxicities, and chronic immune activation/inflammation.

Currently, there is an emerging interest in developing safe and affordable curative strategies that would eliminate the need for lifelong therapy. However, to date only allogeneic hematopoietic stem cell transplantation (allo-HSCT) has shown results in decreasing the HIV-1 reservoirs.

The IciStem Consortium (www.icistem.org) has assembled the largest and most exhaustive observational cohort for the study of HIV reservoir dynamics in allo-HSCT HIV+ individuals with severe hematological malignancies worldwide. Within the cohort, only individuals transplanted with a donor with thw CCR5A32 mutation have shown signs of HIV remission. On the other side broadly neutralizing antibodies (bNAbs) have shown the potential to control HIV infection. This study intends to evaluate if the allo-HSCT combined with the additional application of bNAbs is effective to control HIV replication.

Detailed Description:

The implementation of highly effective, convenient, and well-tolerated combination antiretroviral therapy (cART) for HIV-1 infection has substantially reduced AIDS-related morbidity and mortality. However, cART does not eliminate HIV-1 that persists as a latent infection in cellular reservoirs, including resting memory CD4+ T cells, leading to an underlying raised state of immune activation and subsequent immune senescence. Of note, HIV viremia rapidly rebounds if antiretroviral therapy is interrupted. Consequently, HIV infected individuals must commit to expensive, life-long therapies and must tackle problems associated with chronic infection and uninterrupted cART, including continuous clinical and laboratory monitoring, drug toxicities, and chronic immune activation/inflammation. Therefore, there is an emerging interest in developing safe and affordable curative strategies that would eliminate the need for lifelong therapy while improving the health of infected subjects and reducing the risk of viral transmission to uninfected individuals. So far, allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the only intervention to date that systematically reduces HIV-1 reservoirs to undetectable levels regardless of the CCR5Δ32 donor status.

IciStem is a prospective observational project to investigate cases of allo-HSCT in HIV-1-infected individuals and their putative remission. Over the last few years, the IciStem Consortium (www.icistem.org) has assembled the largest and most exhaustive observational cohort for the study of HIV reservoir dynamics in allo-HSCT HIV+ individuals with severe hematological malignancies worldwide. 39 individuals have already been transplanted and followed up in the IciStem cohort and subsequent undetectable HIV reservoirs in blood and tissues have been described in those with 100% chimerism while still on antiretroviral treatment (ART).

Detailed analysis of CCR5wt allo-HSCT cases within the IciStem cohort has provided insights on additional factors such as conditioning regimen, total body irradiation, graft versus host disease, and viral tropism that contribute to eradication of the potentially infectious viral reservoir in addition to the lack of a functional CCR5 receptor. Allo-HSCT has proved a profound effect on the HIV reservoir. So far, only participants with homozygous CCR5Δ32 mutation have shown signs of HIV remission whereas participants without the CCR5Δ32 mutation had a delayed rebound during ATI. bNAbs have shown the potential to control HIV infection. Consequently, the combination of allo-HSCT with these antibodies is one of the aims of the study by which new cases of HIV remission might be achieved in this setting.

During the last 48 months IciStem has generated a prospective observational cohort of 39 cases of allo-HSCT in HIV-positive participants with severe hematological malignancies in 21 clinical sites in 9 countries (Europe and Canada). Those 39 cases (from the 45 registered) have been followed up with continuous sample collection and high-resolution state of the art virological and immunological analysis. A summary of preliminary studies and achievements is listed below

1. Nine transplants involved CCR5Δ32/Δ32 donors, and 18 involved CCR5wt donors.
2. Mean post-HSCT follow-up is 1656 days, with 18 participants alive in active follow-up (4 transplanted with CCRΔ32/Δ32 donor); 13 IciStem participants are beyond the 2nd year post-HSCT, respectively. From those, 8 are out of immune suppression and with minimal-undetectable HIV latent reservoirs.
3. Five participants from the IciStem Cohort are currently suitable to enter in the first ITATI approach within the IciStem core. Those 5 participants have no detectable replication competent HIV reservoir in presence of cART and have been followed up for the longest time.

The therapeutically intervention for these participants will be an analytical treatment interruption with additional application of broadly neutralizing antibodies (bNAbs) that recently have been described as safe and effective to control HIV replication in infected participants. The rationale for application of these bNAbs during the treatment interruption of the IciStem participants:

* To help prevent viral rebound in absence of cART, due to their proven capacity to potently and durably suppress any possible residual HIV replication
* To rapidly eliminate a cell producing virus via mechanisms such as ADCC (Antibody dependent cellular cytotoxicity)
* To facilitate the development of a broad CTL (Cytotoxic T lymphocytes) response sufficient to maintain remission, as demonstrated in macaques/SHIV studies (Nishimura, 2017)
* To protect the individuals from a putative viral rebound with a safe system, as bNAbs application has few side effects and rarely causes adverse events
* To achieve a highly specific targeting and inhibition of HIV to avoid massive overall bystander activation of the immune system that in effect could lead to a higher chance of HIV reinfection of activated CD4+ T cells.

Despite cART has substantially reduced HIV-related morbidity and mortality, HIV reservoirs are still present and represent a key concern currently for HIV remission. This fact has resulted in a chronicity of HIV infection, leading to emotional disturbances and psychological burden associated with this perpetuation of the disease in the daily living. In the setting of HIV eradication trials, analytical interruption of antiretroviral therapy is a requirement to investigate HIV remission, control, and potential viral rebound. However, discontinuation of cART is linked to psychological issues that should be considered in the setting of HIV cure trials:

1. Stopping cART may lead to variable clinical detriments. Those detriments may induce worry and psychological distress, which can not only worsen the quality of life, but also cause an instability of the emotional status. At the same time, that breakdown of the emotional system may influence the clinical status. Even when clinical consequences are not manifested or self-perceived, beliefs about unfavorable health-related results and desperation for HIV remission may arise.
2. Interrupting cART may increase the risk to infect other people. Those who discontinue cART may not be willing therefore to put their sexual partners at risk. Even after deciding to participate and to interrupt cART, they may develop worries and fears about infecting others.
3. This sort of HIV remission trial comprises a very specific collective of people. People who have suffered from a hematologic medical complication indicative for stem cell transplantation and have survived this severe health problem.

This fact already indicates an impacted emotional status (without even considering the ITATI). Besides, specifically in the current study, additional medical strategies will be applied. Those interventions will be new for the participants (i.e., immune therapy) and will require multiple additional medical appointments. Those characteristics add complexity to the psychological management during the participation in the study.

For all the reasons presented, the participants' psychological predisposition to ITATI and the participation in the study and the emotional status will be monitored carefully throughout the trial. This will be managed at 2 levels: first by continuous assessment of the emotional status and second by offering emotional support whenever required, especially considering the cessation of cART and initiation of the immune therapy.

ELIGIBILITY:
Inclusion Criteria:

* More than 2 years post-HSCT
* Being off immunosuppression for at least one year (related to allo-HSCT)
* Undetectable levels of HIV replication competent reservoirs in blood (< 0,1 IUPM).
* CD4 count levels higher than 200 cel/mm3.
* Aged at least 18 years and not older than 65 at the day of screening
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* In the opinion of the principal investigator or designee, the participant has understood the information provided and capable of giving written informed consent.
* If heterosexually active female; using an effective method of contraception (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner1) from 14 days prior to the first bNAbs administration until at least 6 months after the last bNAbs administration; all female volunteers must be willing to undergo urine pregnancy tests at time points specified.
* If heterosexually active male; willing to use an effective method of contraception (anatomical sterility in self) or agree on the use of an effective method of contraception by his partner(hormonal contraception, intra-uterine device (IUD), or anatomical sterility1 from the day of the first bNAbs administration until 6 months after the last bNAbs administration.
* Willing to accept blood draws at time points specified.
* Not sharing injection drug equipment, such as needles.

  1. Condom use nor diaphragm are considered as an additional method of contraception only and cannot be the only method of contraception used as not been considered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Exclusion Criteria:

* Pregnancy or lactating
* Participation in another clinical trial within 12 weeks of study entry (at screening period).
* History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Time to reappearance of HIV-1 viremia | From Baseline to 18 months
  Time to reappearance of HIV-1 viremia (plasma HIV-1 RNA level > 50 copies/ml in 2 consecutive measurements) after ART interruption.
Time to reappearance of HIV-1 replication competent reservoir | From Baseline to 18 months
  Time to reappearance of HIV-1 replication competent reservoir (determined by the number of infectious units per 106 CD4+ T cells (IUPM) using a viral outgrowth assay) after ART interruption.
Time to reappearance of HIV-1 total reservoir | From Baseline to 18 months
  Time to reappearance of HIV-1 total reservoir (determined by the number HIV-DNA copies per 106 CD4+ T cells using ddPCR) after ART interruption.

SECONDARY OUTCOMES:
Rate and severity of adverse events (AE) and serious adverse events (SAE) | From Baseline to 18 months
  Safety evaluation, as measured by rate and severity of adverse events (AE) and serious adverse events (SAE).
Serum levels of 3BNC117 and 10-1074 | From Baseline to 18 months
  Serum levels of 3BNC117 and 10-1074 throughout the study

OTHER OUTCOMES:
Levels of residual HIV-1 RNA and viral proteins in plasma | Visits from Baseline to 8 months
  Levels of residual HIV-1 RNA and viral proteins in plasma before, during and after infusions of 3BNC117 and 10-1074.
Levels of cellular HIV-1 RNA | Visits from Baseline to 8 months
  Levels of cellular HIV-1 RNA before, during and after infusions of 3BNC117 and 10-1074
Quality of the autologous antibodies. | Visits from Baseline to 8 months
  HIV-1 specific humoral cell immune responses before, during and following 3BNC117 and 10-1074 infusions, including quantity and quality of the autologous antibodies.
Quantity of the autologous antibodies. | Visits from Baseline to 8 months
  HIV-1 specific humoral cell immune responses before, during and following 3BNC117 and 10-1074 infusions, including quantity and quality of the autologous antibodies.
Immunophenotype and functional characteristics of NK, B and T cells from peripheral blood | Visits from Baseline to 8 months
  Immunophenotype and functional characteristics of NK, B and T cells from peripheral blood before, during and following the 3BNC117 and 10-1074 infusions.
Measurement of Immune activation and proliferation markers | Visits from Baseline to 8 months
  Measurement of immune activation and proliferation markers, before, during and following 3BNC117 and 10-1074 infusions.
Measurement of plasma biomarkers | At viral rebound
  Measurement of plasma biomarkers and relate them to HIV viral rebound.
Genome amplification (SGA), phenotypic characterization and full genome analysis of rebounded viruses | From Baseline and 12 weeks after viral re-suppression
  Single genome amplification (SGA), phenotypic characterization and full genome analysis (integration sites and tropism) of rebounded viruses after ART interruption, and after at least 12 weeks after ART re-suppression of viral replication
Immunophenotype and functional characteristics of viral specific T cells | At viral rebound
  Immunophenotype and functional characteristics of viral specific T cells in the viral rebound.
Measurement of HIV-1 total reservoir | At 18 months without viral rebound
  Measurement of HIV-1 total reservoir (determined by the number of HIV-DNA or HIV-RNA copies using ddPCR) in ileum, bone marrow, lymph node and CSF biopsies after 18 months of treatment interruption without viral rebound.
Evaluation of the HIV latent reservoirs in blood | At 18 months without viral rebound
  Evaluation of the HIV latent reservoirs in blood by infusion of the participant's CD4+ T cells in a mice model after 18 months of treatment interruption without viral rebound.
Measurement of ultra-chimerism in blood and tissue populations | Visits from Baseline to 8 months
  Measurement of ultra-chimerism in blood and tissue populations before, during and after the 3BNC117 and 10-1074 infusions
Analysis of metabolic products of glycolysis in plasma | Visits from Baseline to 8 months
  Analysis of metabolic products of glycolysis in plasma before, during and after the 3BNC117 and 10-1074 infusions.
Change in the scores assessing psychological predisposition to Analytical Treatment Interruption (ATI) and emotional status | At Screening, Baseline, 1 month, 8 months, 9 months, 12 months, 18 months and 3 months after viral suppression
  Evaluation of significant change in the scores assessing psychological predisposition to Analytical Treatment Interruption (ATI) and emotional status.
Quantification of the satisfaction level | At 8 months, 18 months and 3 months after viral suppression
  Quantification of the satisfaction levels of the participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Diez, Principal Investigator — Gregorio Marañón Hospital; Manuel Jurado, Principal Investigator — Complejo Hospitalario Universitario de Granada; Alessandra Bandera, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico de Milano; Annemarie Wensing, Principal Investigator — UMC Utrecht
Locations (4):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Lombardy, Italy
- University Medical Center Utrecht, Utrecht, Netherlands
- Spain (2):
  - Complejo Hospitalario Universitario de Granada, Granada, Andalusia
  - Hospital Gregorio Marañón, Madrid